CLINICAL TRIAL: NCT05479812
Title: A Multicenter Phase I/Ib Dose Escalation and Expansion Study of WTX-124 as Monotherapy and in Combination With Pembrolizumab in Patients With Selected Advanced or Metastatic Solid Tumors
Brief Title: Dose Escalation and Expansion Study of WTX-124 as Monotherapy and in Combination With Pembrolizumab (Pembro) in Patients With Selected Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Werewolf Therapeutics, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WTX-124x2101; MK-3475-D17 (Other: Merck Sharp & Dohme LLC); KEYNOTE-D17 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2022-07-14; First posted 2022-07-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Solid Tumor; Advanced Solid Tumor
Keywords: WTX-124; pembrolizumab; Tumors; Cutaneous Malignant Melanoma; mRCC; Renal Carcinoma; IL-2; Cutaneous SCC (cutaneous squamous cell carcinoma); NSCLC (non-small cell lung cancer)
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Melanoma, Cutaneous Malignant; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- WTX-124 monotherapy dose escalation (Experimental): WTX-124 monotherapy dose escalation
  Interventions: Drug: WTX-124
- WTX-124 in combination with pembro dose escalation (Experimental): WTX-124 in combination with pembrolizumab (pembro) dose escalation
  Interventions: Drug: WTX-124; Drug: pembrolizumab
- Arm A: WTX-124 monotherapy dose expansion. Patients with advanced or metastatic RCC. (Experimental): Arm A: WTX-124 monotherapy dose expansion. Patients with advanced or metastatic RCC.
  Interventions: Drug: WTX-124
- Arm B: WTX-124 monotherapy dose expansion. Advanced or metastatic cutaneous malignant melanoma. (Experimental): Arm B: WTX-124 monotherapy dose expansion. Patients with advanced or metastatic cutaneous malignant melanoma.
  Interventions: Drug: WTX-124
- Arm C: WTX-124 monotherapy dose expansion. Patients with advanced or metastatic cSCC. (Experimental): Arm C: WTX-124 monotherapy dose expansion. Patients with advanced or metastatic cSCC.
  Interventions: Drug: WTX-124
- Arm D: WTX-124 in combination with pembro dose expansion. Advanced or metastatic RCC. (Experimental): Arm D: WTX-124 in combination with pembrolizumab dose expansion. Patients with advanced or metastatic RCC.
  Interventions: Drug: WTX-124; Drug: pembrolizumab
- Arm E: WTX-124 with pembro dose expansion. Advanced or metastatic cutaneous melanoma. (Experimental): Arm E: WTX-124 in combination with pembrolizumab dose expansion. Patients with advanced or metastatic cutaneous melanoma.
  Interventions: Drug: WTX-124; Drug: pembrolizumab
- Arm F: WTX-124 in combination with pembro dose expansion. Advanced/metastatic PD-L1-positive NSCL (Experimental): Arm F: WTX-124 in combination with pembrolizumab dose expansion. Patients with advanced or metastatic PD-L1-positive NSCLC lines.
  Interventions: Drug: WTX-124; Drug: pembrolizumab

INTERVENTIONS:
Drug: WTX-124 — Investigation Product Monotherapy
Drug: pembrolizumab — Investigation Product in combination with approved therapy
  Other Names: KEYTRUDA®
  Arms: Arm D: WTX-124 in combination with pembro dose expansion. Advanced or metastatic RCC.; Arm E: WTX-124 with pembro dose expansion. Advanced or metastatic cutaneous melanoma.; Arm F: WTX-124 in combination with pembro dose expansion. Advanced/metastatic PD-L1-positive NSCL; WTX-124 in combination with pembro dose escalation

SUMMARY:
A first-in-human, Phase I, open-label, multicenter study of WTX-124 administered as monotherapy and in combination with pembrolizumab to patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, Phase I, open-label, multicenter study designed to evaluate the safety, tolerability and preliminary efficacy of WTX-124, a conditionally-activated IL-2 prodrug, when administered as monotherapy and in combination with pembrolizumab, for the treatment of patients with advanced solid tumors. Part 1 of the study is dose escalation of WTX-124, both as monotherapy and in combination with pembrolizumab. Part 2 is dose expansion and is comprised of six arms in which WTX-124 will be administered as monotherapy and in combination with pembrolizumab to patients with advanced or metastatic cutaneous malignant melanoma or advanced or metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all the following criteria to participate in the study:

1. Has histological or cytological documentation of a solid tumor indication for which a CPI (e.g. anti-PD-(L)1 is indicated for all parts of the clinical study;
2. Monotherapy Dose Escalation:

   Patients with relapsed/refractory locally advanced or metastatic solid tumors for which immunotherapy is approved, who have progressed on or are intolerant to standard therapy, including CPIs, or for whom no standard therapy with proven benefit exists.

   Combination Dose Escalation:

   Patients with relapsed/refractory locally advanced or metastatic solid tumors for which immunotherapy is approved, who have progressed on or are intolerant to standard therapy or for whom no standard therapy with proven benefit exists.

   Monotherapy Dose Expansion:
   * Arm A: Patients with relapsed advanced or metastatic RCC who have received no more than 4 prior lines of therapy in the advanced or metastatic setting
   * Arm B: Patients with relapsed advanced or metastatic cutaneous malignant melanoma who have received no more than 2 prior lines of therapy for BRAF V600 wild type and no more than 3 prior lines of therapy for BRAF V600 mutant melanoma.
   * Arm C: Patients with relapsed advanced or metastatic cSCC who have received no more than 2 prior lines of systemic therapy

   Combination Dose Expansion:
   1. Arm D: Patients with RCC who have received no more than 3 prior lines of therapy
   2. Arm E: Patients with cutaneous melanoma who may be naïve to all prior therapy for advanced or metastatic disease. For BRAF wild type melanoma, patients should have received no more than 2 prior lines of therapy. For BRAF V600 mutant disease, patients should have received no more than 3 prior lines of therapy.
   3. Arm F: Patients with PD-L1-positive NSCLC who have received no more than 3 prior lines;
3. ≥18 years of age;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
5. Has at least 1 measurable lesion per RECIST 1.1(lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions);
6. Agrees to undergo a pre-treatment and on-treatment biopsy of a primary or metastatic solid tumor lesion;
7. Has adequate organ and bone marrow function;
8. Willingness of men and women of reproductive potential to observe highly effective birth control for the duration of treatment and for 4 months following the last dose of study drug;
9. Additional criteria may apply

Exclusion Criteria:

1. Have a history of another active malignancy (a second cancer) within the previous 2 years except for localized cancers that are not related to the current cancer being treated, are considered cured, and, in the opinion of the Investigator, presents a low risk of recurrence. These exceptions include, but are not limited to, basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast;
2. Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease;
3. Have received prior IL-2-directed therapy;
4. Have had an allogeneic tissue/solid organ transplant;
5. Have known symptomatic brain metastases requiring steroids;
6. Have significant cardiovascular disease;
7. Have an active autoimmune disease that required systemic treatment in the past 2 years;
8. Diagnosis of immunodeficiency, is on immunosuppressive therapy, or is receiving chronic systemic or enteric steroid therapy
9. Major surgery (excluding placement of vascular access) within 2 weeks prior to the first dose of study drug;
10. Investigational agent or anticancer therapy within 5 half-lives or 4 weeks (whichever is shorter) prior to the first dose of study drug;
11. Has received prior radiotherapy within 2 weeks of start of study treatment. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease;
12. Any unresolved toxicities from prior therapy greater than NCI CTCAE version 5.0 Grade 1 at the time of starting study drug with the exception of alopecia and Grade 2 prior platinum-therapy related neuropathy;
13. Received a live or live-attenuated vaccine within 30 days of the first dose of study drug; Note: Administration of killed vaccines or other formats are allowed.
14. Active, uncontrolled systemic bacterial, viral, or fungal infection;
15. HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease;
16. Active infection as determined by hepatitis B surface antigen and hepatitis B core antibody, or hepatitis B virus DNA by quantitative polymerase chain reaction (qPCR) testing;
17. Active infection as determined by hepatitis C virus (HCV) antibody or HCV RNA by qPCR testing;
18. Pregnant or lactating;
19. History of hypersensitivity to any of the study drug components;
20. Additional criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) in monotherapy and combination therapy | 4 weeks
Incidence of treatment emergent adverse events in monotherapy and combination therapy | 24 months
Incidence of changes in clinical laboratory abnormalities in monotherapy and combination therapy | 24 months
Dose Expansion - Incidence of Dose Limiting Toxicities (DLTs) in monotherapy and combination therapy | 4 weeks
Dose Expansion - Incidence of treatment emergent adverse events in monotherapy and combination therapy | 24 months
Dose Expansion - Incidence of changes in clinical laboratory abnormalities in monotherapy and combination therapy | 24 months
Dose Expansion - Investigator-assessed objective response rate (ORR) per RECIST 1.1 and iORR by iRECIST in monotherapy and combination therapy | 24 months

SECONDARY OUTCOMES:
Plasma concentrations of WTX-124 and free IL-2 | 24 months
Investigator-assessed objective response rate (ORR) per RECIST 1.1 and iORR by iRECIST in monotherapy and combination therapy | 24 months
Changes in circulating immune cell populations in response to monotherapy and combination therapy | 24 months
Changes in soluble cytokines in response to monotherapy and combination therapy | 24 months
Changes in tumor immune profile in response to monotherapy and combination therapy | 24 months
Investigator-assessed objective response rate (ORR) per RECIST 1.1 and iORR by iRECIST in monotherapy and combination therapy (in advanced or metastatic renal cell carcinoma and advanced or metastatic cutaneous malignant melanoma) | 24 months
Antidrug antibody (ADA) occurrence | 24 months
Duration of response | 24 months
Progression free survival | 24 months
Overall survival | 36 months
To investigate immunological biomarkers in peripheral blood and tumor that may correlate with the treatment outcome of WTX-124 as monotherapy or in combination with pembrolizumab | 24 months
To assess tumor biopsies for potential biomarkers of target engagement and immune pathway activation | 24 months

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - HonorHealth, Scottsdale, Arizona
  - Moffitt Cancer Center, Tampa, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Minnesota Oncology Hematology, P.A., Maple Grove, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Care, Buffalo, New York
  - Westchester Medical Center, Hawthorne, New York
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Texas Oncology - Austin Midtown, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - NEXT Oncology, Houston, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No